CLINICAL TRIAL: NCT03101280
Title: A Phase IB Combination Study of Rucaparib (CO-338) and Atezolizumab (MPDL3280A) in Participants With Advanced Gynecologic Cancers and Triple-Negative Breast Cancer
Brief Title: A Combination Study of Rucaparib and Atezolizumab in Participants With Advanced Gynecologic Cancers and Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO39409; 2016-002610-47 (EudraCT Number)
Record Dates: First submitted 2017-04-03; First posted 2017-04-05 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Gynecologic Neoplasms
MeSH Terms: conditions — Genital Neoplasms, Female | interventions — atezolizumab; rucaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-Finding Phase (Part 1): Rucaparib and Atezolizumab (Experimental): Approximately 6-18 participants with advanced gynecological cancers will receive different doses of rucaparib administered orally (PO) twice daily (BID) with a fixed dose of atezolizumab (1200 milligrams [mg] intravenously [IV], every 21 days) in 21-day cycles, starting with 400 mg rucaparib BID. The recommended Phase II dose (RP2D), determined by the highest dose level with an acceptable safety profile and with a minimum of 6 participants at which fewer than one-third of participants experience a DLT, was identified as 600 mg rucaparib twice a day (BID).
  Interventions: Drug: Atezolizumab; Drug: Rucaparib
- Dose-Expansion Phase (Part 2): Rucaparib and Atezolizumab (Experimental): Two tumor-specific expansion cohorts will begin treatment with a 21-day run-in period of rucaparib monotherapy at the specified dose for rucaparib in the potential RP2D identified in Part 1 for the combination. Cohort 1 will have approximately 30 participants with advanced, platinum-sensitive ovarian cancer with tumors harboring a tBRCA mutation [tBCRA(mut)] or BRCA-like molecular signature [tBRCA(wt)/LOH(high)].
  Cohort 2 will have approximately 20 participants with previously treated triple-negative breast cancer (TNBC) with a tBRCA mutation [tBCRA(mut)] or BRCA-like molecular signature [tBRCA(wt)/LOH(high)] and have not been exposed to cancer immunotherapies. Following the run in period, participants will receive the combination of rucaparib (specified dose, BID) and atezolizumab (1200 mg IV, every 21 days) in 21-day cycles.
  Interventions: Drug: Atezolizumab; Drug: Rucaparib

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg (equivalent to an average body weight-based dose of 15 milligrams per kilogram [mg/kg]) will be administered by IV infusion once every 3 weeks, corresponding to a 21-day treatment cycle. Participants will receive atezolizumab starting on Cycle 1, Day 1. Participants deriving clinical benefit will be allowed to continue on study treatment until the absence of unacceptable toxicity or compelling evidence of disease progression.
  Other Names: MPDL3280A; TECENTRIQ
Drug: Rucaparib — The starting dosage level of rucaparib for Part 1 is 400 mg PO BID during a 21-day treatment cycle. During Part 1, the rucaparib doses were increased up to a maximum of 600 mg PO BID using a standard 3 + 3 dose escalation. RP2D was identified as 600 mg BID. During Part 2 of the study, rucaparib will be dosed at the RP2D determined in Part 1. Participants in Part 1 of the study will receive rucaparib starting on Cycle 1, Day 1. During Part 2, participants will receive rucaparib monotherapy during a 21-day run-in period. After completion of the rucaparib run-in period and the first on-treatment biopsy between Days 15 and 21 of the run-in period, participants will begin Cycle 1, Day 1 of the rucaparib. Participants deriving clinical benefit will be allowed to continue on study treatment until the absence of unacceptable toxicity or compelling evidence of disease progression.
  Other Names: CO-338

SUMMARY:
This is a Phase Ib, open-label, non-randomized study in patients with previously treated advanced ovarian or endometrial cancer (Part 1) and platinum-sensitive ovarian cancer or triple-negative breast cancer (TNBC) (Part 2) to investigate the dose, safety, pharmacokinetics, and preliminary efficacy of rucaparib in combination with atezolizumab. The study is conducted in 2 parts: a Dose-Finding Phase (Part 1) and a Dose-Expansion Phase (Part 2)

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* A life expectancy of at least 3 months
* Have disease that is measurable as according to RECIST v1.1
* Have sufficient archival formalin-fixed paraffin-embedded (FFPE) tumor tissue available for planned analyses
* For Part 1, have a histologically confirmed diagnosis of ovarian or endometrial cancer, and have received at least one line of prior therapy for metastatic disease
* For Part 2 ONLY, have disease that can be safely biopsied
* For Part 2 ONLY, have a deleterious germline or somatic breast cancer susceptibility gene 1 (BRCA1) or BRCA2 mutation or tumors that are wild-type BRCA but show high levels of loss of heterozygosity (LOH) (tBRCAwt/LOHhigh) signature
* For Part 2 Cohort 1 (ovarian cancer), high-grade serous or Grade 3 endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer (PPC)
* For Part 2 Cohort 1, have received at least one and no more than two lines of prior platinum-containing therapy and progressed after the most recent platinum therapy in a platinum-sensitive timeframe
* For Part 2 ONLY, Cohort 1, have a CA125 measurement that is greater than 2 times the upper limit of normal (ULN)
* For Part 2 Cohort 2 (TNBC), metastatic, histologically confirmed estrogen receptor (ER)-negative, progesterone receptor-negative, and HER2-negative adenocarcinoma of the breast per local laboratory assessment
* For Part 2 Cohort 2, radiologic/objective evidence of recurrence or disease progression after one line of chemotherapy for TNBC in the metastatic setting
* Have adequate organ function

Exclusion Criteria:

* History of prior malignancy except a) curatively treated non-melanoma skin cancer, b) solid tumor treated curatively more than 3 years ago without evidence of recurrence, c) For Cohort 1 (ovarian cancer): breast cancer with no evidence of disease or inactive for at least 3 years, and d) synchronous endometrial cancer (Stage 1A) with ovarian cancer
* Treatment with chemotherapy, radiation, hormones (except corticosteroids and megestrol acetate), or other anticancer therapies less than or equal to (<=) 14 days prior to first dose of study treatment
* Preexisting duodenal stent and/or any gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with absorption of rucaparib
* Symptomatic and/or untreated central nervous system metastases
* Prior treatment with any poly adenosine diphosphate-ribose polymerase (PARP) inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Baseline up to approximately 45 months
Percentage of Participants With Dose-Limiting Toxicities (DLTs) [Part 1] | Cycle 1 (Day 1 up to Day 21)
Recommended Phase II Dose (RP2D) of Rucaparib for the Combination [Part 1] | Cycle 1 (Day 1 up to Day 21)
Number of Dose Modifications due to Adverse Events [Part 2] | Baseline up to approximately 45 months

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response of Complete Response (CR) or Partial Response (PR) as Determined by Investigator Assessment Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Baseline until disease progression or death from any cause, whichever occurs first (assessed every 12 weeks up to approximately 45 months)
Percentage of Participants With Objective Response of CR or PR as Determined by Investigator Assessment Using Immune-Modified RECIST Incorporating Immune-Response (Cancer Antigen 125 [CA125] Response) Considerations | Baseline until disease progression or death from any cause, whichever occurs first (assessed every 12 weeks up to approximately 45 months)
Duration of Response (DOR) as Determined by Investigator Assessment Using RECIST v1.1 | Baseline until disease progression or death from any cause, whichever occurs first (assessed every 12 weeks up to approximately 45 months)
DOR as Determined by Investigator Assessment Using Immune-Modified RECIST Incorporating Immune-Response (CA125 Response) Considerations | Baseline until disease progression or death from any cause, whichever occurs first (assessed every 12 weeks up to approximately 45 months)
Progression-Free Survival (PFS) as Determined by Investigator Assessment Using RECIST v1.1 | Baseline until disease progression or death from any cause, whichever occurs first (assessed every 12 weeks up to approximately 45 months)
PFS as Determined by Investigator Assessment Using Immune-Modified RECIST Incorporating Immune-Response (CA125 Response) Considerations | Baseline until disease progression or death from any cause, whichever occurs first (assessed every 12 weeks up to approximately 45 months)
Overall Survival | Baseline until Death (up to 45 months)
Steady State Maximum Plasma Concentration Observed (Cmax) for Rucaparib [Part 1] | Predose (0 hours [hrs]) on Day 1 of Cycles 1-4; 0, 0.5, 1, 1.5, 2.5, 4, 6, 8 hrs postdose on Day 15 of Cycle 1; at 30 days after the last dose of study treatment (up to 45 months; cycle length=21 days)
Time to Maximum Plasma Concentration (tmax) for Rucaparib [Part 1] | Predose (0 hrs) on Day 1 of Cycles 1-4; 0, 0.5, 1, 1.5, 2.5, 4, 6, 8 hrs postdose on Day 15 of Cycle 1; at 30 days after the last dose of study treatment (up to 45 months; cycle length=21 days)
Area Under the Plasma Concentration-Time Curve (AUC) for Rucaparib [Part 1] | Predose (0 hrs) on Day 1 of Cycles 1-4; 0, 0.5, 1, 1.5, 2.5, 4, 6, 8 hrs postdose on Day 15 of Cycle 1; at 30 days after the last dose of study treatment (up to 45 months; cycle length=21 days)
Apparent Clearance (CL/F) for Rucaparib [Part 1] | Predose (0 hrs) on Day 1 of Cycles 1-4; 0, 0.5, 1, 1.5, 2.5, 4, 6, 8 hrs postdose on Day 15 of Cycle 1; at 30 days after the last dose of study treatment (up to 45 months; cycle length=21 days)
Minimum Plasma Concentration During the Dosing Interval (Cmin) for Rucaparib [Part 2] | Predose (0 hrs) on Day 1 of Cycles 1-4; at 30 days after the last dose of study treatment (up to 45 months; cycle length=21 days)
Serum Concentration of Atezolizumab [Parts 1 and 2] | Predose (0 hrs) on Day 1 of Cycles 1-4, 8 and every 8 cycles (up to 45 months); 0.5 hrs postdose (infusion duration=30-60 minutes) on Day 1 of Cycles 1 and 3; at 30 and 120 days after last dose of study treatment (up to 45 months; cycle length=21 days)
Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab | Baseline up to approximately 45 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Peter Maccallum Cancer Centre, Melbourne, Victoria, Australia
- France (3):
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Lyon Sud; Service d'Oncologie Médicale, Pierre-Bénite
  - Gustave Roussy, Villejuif
- Spain (3):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron, Barcelona
  - La Paz University Hospital, Madrid
- United Kingdom (4):
  - Royal Marsden Hospital - London, London
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Kristeleit R, Leary A, Oaknin A, Redondo A, George A, Chui S, Seiller A, Liste-Hermoso M, Willis J, Shemesh CS, Xiao J, Lin KK, Molinero L, Guan Y, Ray-Coquard I, Mileshkin L. PARP inhibition with rucaparib alone followed by combination with atezolizumab: Phase Ib COUPLET clinical study in advanced gynaecological and triple-negative breast cancers. Br J Cancer. 2024 Sep;131(5):820-831. doi: 10.1038/s41416-024-02776-7. Epub 2024 Jul 6. PMID 38971950